CLINICAL TRIAL: NCT03957759
Title: Self-Monitoring for Early Signs of Altitude Illness in Patients With Chronic Obstructive Pulmonary Disease. A Diagnostic Test Accuracy Study.
Brief Title: Early Signs of Altitude Illness in Patients With COPD
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01-8/464-14
Record Dates: First submitted 2019-05-16; First posted 2019-05-21 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Altitude; Hypobaric hypoxia; Altitude-related illness; Prevention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients
  Interventions: Diagnostic Test: Structured self-monitoring during an altitude ascent and stay at high altitude

INTERVENTIONS:
Diagnostic Test: Structured self-monitoring during an altitude ascent and stay at high altitude — Structured self-monitoring by a symptom checklist in combination with a pulse oximeter worn at the wrist in lowlanders with COPD ascending from low altitude (760m) to high altitude (3100m).

SUMMARY:
This study evaluates whether structured self-monitoring (SSM) by a symptom checklist in combination with a pulse oximeter worn at the wrist allows lowlanders with COPD to accurately identify whether or not they will experience an altitude-related illness during altitude travel.

DETAILED DESCRIPTION:
This study evaluates whether structured self-monitoring (SSM) by a symptom checklist in combination with a pulse oximeter worn at the wrist allows lowlanders with COPD to accurately identify whether or not they will experience an altitude-related illness during altitude travel. After baseline evaluation at 760 m, patients will travel by bus within 3-5 h to the Tuja Ashu high altitude clinic at 3'100 m and stay there for 2 days. During this period, participants will perform SSM. They are instructed to report to study personnel if they fulfill predefined criteria for impeding altitude-related illness.

A planned interim analysis will be performed after the first year of the study or after completion of study by 80 participants, whichever comes first to allow any necessary adaptations of the sample size or terminate the study early for futility or high accuracy of the index test.

ELIGIBILITY:
Inclusion criteria

* Male and female patients, age 18-75 yrs.
* COPD diagnosed according to GOLD, FEV1 40-80% predicted, SpO2 ≥92%, PaCO2 <6 kPa at 760 m.
* Born, raised and currently living at low altitude (<800 m).
* Written informed consent.

Exclusion criteria

* COPD exacerbation, very severe COPD with hypoxemia at low altitude (FEV1 <40% predicted; oxygen saturation on room air <92% or hypercapnia at 760 m).
* Other lung disease or disorder of control of breathing
* Comorbidities such as uncontrolled cardiovascular disease, i.e., unstable systemic arterial hypertension, coronary artery disease; previous stroke, internal, neurologic, rheumatologic or psychiatric disease that interfere with protocol compliance including current heavy smoking (>20 cigarettes per day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD, FEV1 40-80% predicted living at low altitude.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic accurarcy measures of structured self-monitoring | Day 1 to 3 at 3100m
  Diagnostic performance includes sensitivity, specificity, positive and negative predictive values, and receiver operator curve area under the the curve. The diagnostic performance will be compared statistically using c-statistics against the reference test. Reference test will be the occurence of altitude-related illness defined as the following:
  * AMS defined by the Lake Louise questionnaire score or with AMSc score
  * severe hypoxemia (SpO2 <80% at rest >30 min; or SpO2 <75% at rest >15 min;
  * intercurrent illness that cannot be relieved by simple measures such as paracetamol 3x500 mg/day, inhalation of bronchodilators.
  * dyspnea or discomfort at rest requiring treatment with oxygen
  * chest pain or ECG signs of cardiac ischemia
  * severe hypertension: systolic blood pressure >200 mmHg, diastolic blood pressure >110 mmHg
  * new onset neurologic impairment
  * Any condition that requires study withdrawal according to the decision of the independent physician

SECONDARY OUTCOMES:
Acute mountain sickness severity assessed by the Lake Louise score | Day 1 to 3 at 3100m
  The severity of acute mountain sickness will be assessed by the Lake Louise questionnaire. The severity will be calculated when the presence of headache and at least one of the following symptoms is present: gastrointestinal upset, fatigue or weakness and dizziness or lightheadedness. Each of the four questions is asked with the corresponding 0 to 3 rating of the response (0 = Not present, 1 = mild, 2 = moderate, 3 = severe). The sum of the responses on these questions is then calculated, resulting in the AMS severity.
Altitude-related illness, incidence | Day 1 to 3 at 3100m
  Incidence of ARI during the stay at 3100 m.
  ARI is defined as the following:
  * AMS defined by the Lake Louise questionnaire score or with AMSc score
  * severe hypoxemia (SpO2 <80% at rest >30 min; or SpO2 <75% at rest >15 min;
  * intercurrent illness that cannot be relieved by simple measures such as paracetamol 3x500 mg/day, inhalation of bronchodilators.
  * dyspnea or discomfort at rest requiring treatment with oxygen
  * chest pain or ECG signs of cardiac ischemia
  * severe hypertension: systolic blood pressure >200 mmHg, diastolic blood pressure >110 mmHg
  * new onset neurologic impairment
  * Any condition that requires study withdrawal according to the decision of the independent physician
Spirometric measurement of forced expiratory volume in one second | Day 2 at 760 and 3100m
  Altitude-induced change in the forced expiratory volume in one between 760 and 3100m
Arterial partial pressure of oxygen | Day 2 at 760 and 3100m
  Altitude-induced change in arterial partial pressure of oxygen assessed by arterial blood gas puncture at 760 and 3100m
Six-minute walk distance in meters | Day 2 at 760 and 3100m
  Altitude-induced change in the six-minute walk distance assessed by the six-minute walk test performed at 760 and 3100m
Changes in ST-Segment of the ECG during ergometry | Day 1 at 760 and 3100m
  Altitude-induced change in the ST-Segment of the ECG assessed during a maximal ergometry test performed at 760 and 3100m

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University of Zurich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

REFERENCES:
- [Derived] Furian M, Reiser AE, Mademilov M, Sutter S, Champigneulle B, Grimm M, Magdieva K, Beishenaliev AS, Sooronbaev TM, Ulrich S, Bloch KE. Self-monitoring symptoms and pulse oximetry to predict imminent altitude illness in patients with chronic obstructive pulmonary disease. Pulmonology. 2026 Dec;32(1):2588515. doi: 10.1080/25310429.2025.2588515. Epub 2025 Dec 23. PMID 41433778